CLINICAL TRIAL: NCT02789995
Title: Dysfunctions of Human Muscle Stem Cells in Sepsis
Acronym: DISCUSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-015; ID-RCB number : 2015-A01022-47 (Other: French national registration number of the study)
Record Dates: First submitted 2016-05-18; First posted 2016-06-03 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Sepsis
Keywords: Intensive Care Unit - Acquired Weakness (ICU-AW)
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with and without sepsis (Experimental): Patients with sepsis, Patients with inflammatory disease without sepsis, Patients without inflammatory disease without sepsis.
  Human biological samples collected for research :
  * Blood sample
  * Muscle biopsy
  * Bone marrow sample (mesenchymal stem cells)
  Interventions: Procedure: Human biological samples

INTERVENTIONS:
Procedure: Human biological samples — Blood sample - Muscle biopsy - Bone marrow sample (mesenchymal stem cells)

SUMMARY:
Severe critical illness is often complicated by Intensive Care Unit - Acquired Weakness (ICU-AW), which is associated with increased in and post-ICU mortality, with delayed weaning from mechanical ventilation and with long-term functional. Several mechanisms have been incriminated in the pathophysiology of ICU-AW, but muscle regeneration has not been well investigated in this context, even though its involvement is suggested by the protracted functional consequences of ICU-AW. Recent data suggest that muscle regeneration could be impaired after sepsis, and that Mesenchymal Stem Cells (MSCs) treatment could improve the post-injury muscle recovery.

DETAILED DESCRIPTION:
Severe critical illness is often complicated by Intensive Care Unit - Acquired Weakness (ICU-AW), which is clinically characterized by bilateral and symmetrical limb weakness and is related to a myopathy and/or axonal polyneuropathy. ICU-AW affects between 25% to 60% mechanically ventilated patients more than 7 days and is associated with increased in and post-ICU mortality, with delayed weaning from mechanical ventilation and with long-term functional disability. Most patients who develop an ICU-AW have been admitted for a sepsis episode and the main risk factors of ICU-AW include the severity of critical illness, immobilization, hyperglycemia and the use of some medications including steroids and neuromuscular agents, although this is somewhat controversial.

The pathophysiology of critical illness myopathy is thought to involve the following mechanisms: 1) impairment of muscular membrane excitability, secondary to an dysregulation of sodium channel gating, 2) mitochondrial dysfunction leading to bioenergetic failure and oxidative stress and 3) proteolysis, mainly related an activation of the ubiquitin-proteasome pathway. These mechanisms can be triggered by various factors, notably systemic inflammatory mediators, endocrine dysfunction, immobilization, some drugs and electrolyte disturbances. The protracted functional consequences of ICU-AW indicate that muscle regeneration is also impaired. Surprisingly, muscle regeneration, which essentially depends on the muscle stem cells (also called satellite cells), has not been well investigated in the context of critical illness. The satellite cells (SC), that are located at the periphery of the muscle fiber, are activated in response to any muscle injury and then proliferate and differentiate to repair or replace the damaged fibers, but also self-renew to replenish the muscle stem cells reservoir.

It was recently demonstrated in a murine model of polymicrobial peritonitis that SC activation, proliferation and expression of myogenic markers were impaired after sepsis, leading to an impaired muscle regeneration, but that post-sepsis intramuscular administration of exogenous Mesenchymal Stem Cells (MSCs) could reverse this SC dysfunction. MSC treatment significantly improved the post-injury muscle recovery with decreasing necrosis and fibrosis but also increased the force of isolated single fibers.

The objectives of this translational research are to identify the mechanisms of Human SC dysfunction in patients with severe sepsis, to describe in vitro the effects of MSCs on this SC dysfunction, and to study hematopoietic cells and their damage in the blood and muscle consecutively to a sepsis, and their interaction with muscle stem cells.

ELIGIBILITY:
Inclusion Criteria:

* Affiliated or beneficiary of a social security system
* Informed consent to research :

Consent from patient, Or consent from patient and close relative, Or non-objection from family for biological sample donation for research.

* Population 1 (sepsis) : Patients hospitalized in Intensive Care Unit, with intra-abdominal sepsis requiring emergency surgery.
* Population 2 (inflammatory condition with or without sepsis) : Brain dead patients scheduled for multi organ retrieval (2a) ; Patients with refractory cariogenic shock and requiring surgery for assistance with (2b).
* Population 3 (control) : Patients scheduled for intra-abdominal surgery.

Exclusion Criteria:

* Patient with preexisting neuromuscular disease
* Under 18 year-old
* Pregnancy..

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2016-06-23 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Muscle regenerative capacities | 3 years
  The muscle regenerative capacity after sepsis would be assessed by the presence of anisocytosis, the proportion of small atrophic fibers, the proportion of endomysial fibrosis of the total muscle section area and the presence of calcified necrotic myofibers.

SECONDARY OUTCOMES:
Satellite cell dysfunction after sepsis | 3 years
  * Number of satellite cells (SC)
  * Proportion of cells actively cycling
  * Capacity of SC to differentiate into myofibers
Regenerative capacities of Human satellite cells in presence of mesenchymal stem cells | 3 years
  * Number of satellite cells (SC)
  * Proportion of cells actively cycling
  * Capacity of SC to differentiate into myofibers

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Chrétien, Study Director — Institut Pasteur
Locations (7):
- France (7):
  - Hopital Henri Mondor, Service de Réanimation chirurgicale polyvalente, Créteil
  - Hôpital Pitié Salpétrière, Salle de surveillance post-interventionnelle, Accueil des Polytraumatisés, Paris
  - Hôpital Pitié Salpêtrière, Anesthésie et Réanimation, Institut de Cardiologie, Paris
  - Hôpital Pitié Salpêtrière, Service de Chirurgie Générale, Viscérale et Endocrinienne, Paris
  - Hôpital Pitié Salpêtrière, Service de Chirurgie Hépatobiliaire et de Transplantation Hépatique, Paris
  - Hôpital Pitié Salpêtrière, Service de réanimation chirurgicale polyvalente, Paris
  - Hôpital Saint-Antoine, Département d'Anesthésie-réanimation, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rocheteau P, Chatre L, Briand D, Mebarki M, Jouvion G, Bardon J, Crochemore C, Serrani P, Lecci PP, Latil M, Matot B, Carlier PG, Latronico N, Huchet C, Lafoux A, Sharshar T, Ricchetti M, Chretien F. Sepsis induces long-term metabolic and mitochondrial muscle stem cell dysfunction amenable by mesenchymal stem cell therapy. Nat Commun. 2015 Dec 15;6:10145. doi: 10.1038/ncomms10145. PMID 26666572
- [Derived] Duceau B, Blatzer M, Bardon J, Chaze T, Giai Gianetto Q, Castelli F, Fenaille F, Duarte L, Lescot T, Tresallet C, Riou B, Matondo M, Langeron O, Rocheteau P, Chretien F, Bougle A. Using a multiomics approach to unravel a septic shock specific signature in skeletal muscle. Sci Rep. 2022 Nov 5;12(1):18776. doi: 10.1038/s41598-022-23544-8. PMID 36335235